CLINICAL TRIAL: NCT04698525
Title: Efficacy of Memantine Compared With Sodium Valproate in the Prophylactic Treatment of Episodic Migraine.
Brief Title: Comparative Study Between Valproate and Memantine in the Prophylactic Management of Episodic Migraine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Ildefonso Rodriguez-Leyva, MD, PhD, FAAN, FANA, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 74-19
Record Dates: First submitted 2020-12-08; First posted 2021-01-07 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Migraine Headache
Keywords: Episodic MIgraine; Memantine; Valproate; Efficacy; Security; MIDAS; Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — Valproic Acid; Memantine

STUDY DESIGN:
Intervention Model Description: A double-blind study with two groups. One using VPA and the other one using memantine in subjects with a diagnosis of episodic migraine.
Who Masked: Investigator
Masking Description: The clinician will make an evaluation and if the patient has the criteria for inclusion will be by randomization in one group or another. Neither the clinician and the patient will not know the administrated treatment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Valproate group (Active Comparator): This is a well know antiepileptic drug with efficacy as a preventive tic treatment in episodic migraine
  Interventions: Drug: Valproate Sodium
- Memantine (Active Comparator): This is a possible preventive treatment in episodic migraine
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Valproate Sodium — Comparison between two actives
  Other Names: Diwali
  Arms: Valproate group
Drug: Memantine — Memantine
  Other Names: Ezagun
  Arms: Memantine

SUMMARY:
Migraine is one of the three most disabling diseases worldwide. Constituted by recurrent episodes of headache, characterized by unilateral location, throbbing character, moderate or severe intensity, worsening with physical activity, and association with nausea or photophobia and/or phonophobia. There are two types of drug treatment: abortifacient and prophylactic. The American Academy of Neurology classifies sodium valproate as level A; however, some patients do not obtain a satisfactory response rate and/or have adverse effects. Therefore, the search for new pharmacological treatments continues. In 2015, a double-blind, randomized clinical trial with a placebo was carried out to assess Memantine's efficacy in the prophylactic treatment of migraine without aura, which reported a reduction of 2.3 migraine attacks per month compared to the placebo group. Memantine could be a new effective treatment alternative, which is why we will compare the efficacy of Memantine against sodium valproate as a prophylactic migraine treatment.

Main objective: To compare the efficacy of Memantine at a rate of 20mg divided into two doses a day against sodium valproate (VPA) at a rate of 1000mg divided into two doses a day prophylactic treatment of migraine for three months.

Study design: a prospective controlled, randomized, double-blind clinical trial. Inclusion criteria: Men and women aged 18 to 65 years with a diagnosis at least one year before the study must present at least 2 to 8 migraine attacks per month and less than 15 days with headache per month, which should not be receiving prophylactic treatment for migraine and sign an informed consent

Sample size calculation and statistical analysis:

It is calculated using the normal distribution model, where the recommended sample size is 196 participants. Since a pilot study will be conducted, 10% of the sample size will be taken to make it representative, a sample size of 20 participants is decided for each group.

DETAILED DESCRIPTION:
Migraine is a primary headache, currently one of the three most disabling diseases globally. It has an annual and lifetime prevalence of 18% and 33% in women, and 6 to 13% in men, respectively, with a predominance in women (3: 1). The age of onset with the highest prevalence is between 25 and 55 years.

Migraine is described by the International Headache Society (IHS) as recurrent episodes of headache lasting 4 to 72 hours, characterized by unilateral location, pulsatile character, moderate or severe intensity, worsening with physical activity, and association with nausea or photophobia and phonophobia. The IHS also classifies migraine based on the frequency of attacks: episodic migraine when the headache occurs on less than 15 days a month, and chronic migraine, when the headache occurs 15 or more days a month for three months and at least eight days a month with characteristics of migraine headache.

The subtypes of migraine concerning their clinical presentation are migraine with aura and without aura.4 Up to one-third of patients present migraine aura, with visual symptoms being the most frequent.

Four phases have been identified during a migraine: prodromal phase, aura, headache, and postdrome. The prodromal phase is characterized by premonitory symptoms hours before the headache, including difficulty concentrating, irritability, fatigue, repetitive yawning, stiff neck, and photophobia.

Recurrent episodes characterize the aura, lasting from 5min to 60min, with transient unilateral visual, sensory, or other CNS symptoms that develop progressively, usually precede headache and symptoms associated with migraine.4 The aura's genesis is activated by the NMDA (N-methyl-D-aspartate) receptor and disseminated cortical depression. Disseminated cortical depression is an extreme depolarization of the cell membranes of the glia and neurons that produce an alteration of the ionic gradient, an increase in extracellular potassium concentrations, glutamate release, and a transient increase followed by a decrease in cerebral blood flow.

The pain phase in migraine is due to the activation and sensitization of the trigeminovascular pain pathway, which innervates intracranial structures, including the eye, the dura mater, large braincases, and the venous sinuses. It has been shown to involve neuronal presynaptic activation by ID serotonin receptors (5-HT 1D), resulting in the release of the calcitonin gene (CGRP) and pituitary adenylate cyclase-activating polypeptide (PACAP-38), which are neuroinflammatory peptides. The post-synaptic effect on the meninges includes the activation of the arachidonic acid cascade, which conditions inflammation and vasodilation, stimulates the nociceptive afference of pain first branch of the trigeminal nerve.

The diagnosis of migraine is clinical and must meet the criteria of the IHS International Classification of Headaches (ICH-3), which are for migraine without aura:

At least five crises that meet criteria B-D. A. Headache episodes are lasting 4 to 72 hours (untreated or unsuccessfully treated).

B. The headache has at least two of the following four characteristics:

1. Unilateral location.
2. Pulsatile character.
3. Pain of moderate or severe intensity.
4. Made worse by or conditions the abandonment of habitual physical activity (e.g., walking or climbing stairs).

C. At least one of the following during the headache:

1. Nausea and vomiting.
2. Photophobia and phonophobia. D. No better explanation by another diagnosis of ICHD-III.

The non-pharmacological treatment of migraine goes hand in hand with the pharmacological one; one is to avoid the triggers of the migraine attacks and carry out the lifestyle modifications. Pharmacological treatment is divided into acute (administered at the time of headache) and prophylactic (administered daily to reduce the chances of migraine episodes).

The objective of prophylactic treatment is to reduce the frequency, duration, and severity of migraine attacks, improve the response to acute treatment, improve functionality, and reduce disability.

The American Academy of Neurology recommends initiating prophylactic treatment in patients with migraine with one or more of the following characteristics9

1. Recurrent migraine, which interferes with the patient's daily life and quality of life.
2. Frequent headaches.
3. That they have an inadequate response or contraindication to abortive treatment.
4. Adverse events to abortion treatment.
5. Uncommon migraine conditions: ophthalmoplegic migraine, basilar migraine, hemiplegic, prolonged aura, migraine infarction.

The IHS defines the response to treatment as a decrease equal to or greater than 50% in the frequency of migraine attacks compared to the baseline situation.

The American Academy of Neurology guideline for the prophylactic drug treatment of episodic migraine classifies divalproex sodium, valproate sodium (VPA), topiramate, metoprolol propranolol as level A (Drugs with established efficacy ).

Valproic acid (2-propylpentaenoic acid) was first synthesized in 1882 as an analog of valeric acid, naturally found in valerian. Anyone of Valproic acid, sodium valproate, or a mixture of the two (sodium valproate) has a mechanism of action characterized by increasing or improving GABA neurotransmission, blocking voltage-gated sodium channels, and T-type calcium channels. In 2013, Cochrane conducted the review: Valproate for the prophylaxis of episodic migraine (Linda et al.), where they evaluated ten clinical trials. Two crossover clinical trials for sodium valproate demonstrated a significant reduction in headache frequency than placebo (MD -4.31 95% CI -8.32 to -0.30), which shows us in clinical terms an approximate reduction of four headaches for every 28 days. Jensen 199413 showed that sodium valproate is superior to placebo (OR 4.67; 95% CI 1.54 - 14.14), suggesting that patients are three times more likely to present a reduction equal to or greater than 50% in the frequency of headaches compared to placebo. The recommended dose for migraine headaches is 500-1000mg per day. The most common adverse effects are asthenia, fatigue, dizziness/vertigo, nausea, tremor, and weight gain.

In recent years, interest has increased in glutamate receptor antagonists for migraine prophylaxis, such as memantine. Within the pathophysiology of migraine, glutamate is implicated in disseminated cortical depression, trigeminal-vascular activation. Other studies corroborate its role by reporting elevated glutamate levels in the cerebrospinal fluid in patients with chronic migraine in the ictal period and elevated serum levels in migraine patients. Besides, after experimental stimulation in the dura and the ventral-posteromedial thalamic nucleus structures, elevated levels of glutamate in the trigeminal-cervical complex have been evidenced. fifteen

In 2008 Bigal and colleagues conducted the first open clinical trial, a pilot study to evaluate memantine's efficacy and safety as a prophylactic treatment in patients diagnosed with refractory migraine. A sample of 28 participants who had a baseline frequency of headache days of 21.8 days per month received memantine from 10mg to 20mg per day for three months. A decrease in the frequency of headache days was obtained to 16.1 (P <0.01). Therefore, the authors concluded that memantine as a prophylactic treatment is safe and effective in refractory migraines. In 2015, Noruzzadeh and colleagues conducted the first randomized, double-blind, placebo-controlled clinical trial to evaluate memantine's efficacy as a prophylactic treatment of migraine without aura With a sample of 52 participants, 25 with memantine (10 mg/day) and 27 with placebo. The memantine group had a more significant reduction in the frequency of migraine attacks compared to placebo, which was a difference of 2.3 attacks per month with a P <0.001.14

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 to 65 years old.
2. Diagnosis of migraine according to the ICHD-III of the IHS at least one year before the study.
3. You must have at least 4-14 migraine attacks per month.
4. Not receiving prophylactic treatment for migraine
5. Sign informed consent

Exclusion Criteria:

1. Pregnant or lactating patients.
2. Patients with another type of non-migraine headache.
3. Allergy to Sodium Valproate and/or Memantine
4. Being a carrier of systemic disease (infectious, immunological, or metabolic processes) or cardiovascular (myocardial, coronary, or valvular disease) prevents their participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan M. Shiguetomi-Medina, MD, PhD, Study Chair — Facultad de Medicina, Universidad Autonoma de San Luis Potosi
Locations (1):
- Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
This clinical trial is the thesis to obtain a specialist degree (Neurologist) of Dr. Damaris Daniela Vazquez-Guevara; at the end of the study, the plan is to publish as soon as possible.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: 6 months

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Bille B. A 40-year follow-up of school children with migraine. Cephalalgia. 1997 Jun;17(4):488-91; discussion 487. doi: 10.1046/j.1468-2982.1997.1704488.x. PMID 9209767
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Schwedt TJ. Preventive Therapy of Migraine. Continuum (Minneap Minn). 2018 Aug;24(4, Headache):1052-1065. doi: 10.1212/CON.0000000000000635. PMID 30074549
- [Background] Linde M, Mulleners WM, Chronicle EP, McCrory DC. Valproate (valproic acid or sodium valproate or a combination of the two) for the prophylaxis of episodic migraine in adults. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD010611. doi: 10.1002/14651858.CD010611. PMID 23797677
- [Background] Noruzzadeh R, Modabbernia A, Aghamollaii V, Ghaffarpour M, Harirchian MH, Salahi S, Nikbakht N, Noruzi N, Tafakhori A. Memantine for Prophylactic Treatment of Migraine Without Aura: A Randomized Double-Blind Placebo-Controlled Study. Headache. 2016 Jan;56(1):95-103. doi: 10.1111/head.12732. Epub 2015 Dec 6. PMID 26638119

RESULTS

PARTICIPANT FLOW:
Groups:
- Valproate Group: VPA is a well know antiepileptic drug with efficacy as a preventive tic treatment in episodic migraine.
  Valproate Sodium: Comparison between two actives
  There were 17 patients in the valproate group. In both grupus, females represent the majority.
- Memantine: This is a possible preventive treatment for episodic migraine
  Memantine: MemantineThere was 16 patients in the memantine group
Period: Overall Study
Arm/Group | Valproate Group | Memantine
Started | 17 | 16
Completed | 14 | 13
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Three suffered of Covid-19 | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total of 33 subjects participated in the trial, 6 of which left due to covid-19 infections. In the end, 27 subjects completed the trial.
Groups:
- Valproate Group: VPA is a well know antiepileptic drug with efficacy as a preventive treatment for episodic migraine.
  Valproate Sodium
- Total: Total of all reporting groups
Arm/Group | Valproate Group | Memantine | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants] — All the participants were between 18 to 65 years old.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 16 | 33
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.58 (7.51) | 31.18 (10.94) | 31.38 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 17 | 16 | 33
Pain Localization: hemicranial [Count of Participants; unit: Participants] — Subjects with pain on the left or right side of the head only (unilateral) were classified as having Hemicraneal pain. Subjects with pain in both sides of the head were classified as having Holocranial pain.
  Participants
    Hemicraneal pain | 13 | 14 | 27
    Holocranial pain | 4 | 2 | 6
Photophobia [Count of Participants; unit: Participants] | 16 | 14 | 30
Sonophobia [Count of Participants; unit: Participants] | 10 | 16 | 26
Nausea and vomit [Count of Participants; unit: Participants] | 17 | 14 | 31
Disability [Count of Participants; unit: Participants] | 17 | 14 | 31
With aura [Count of Participants; unit: Participants] | 13 | 13 | 26
Without aura [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Days of Headache Pain With Treatment of Memantine or Valproate in the Preventive Management of Episodic Migraine.
Description: In a double-blind clinical trial, we compared two active drugs (mamantine vs. valproate) three months after initiation, looking for changes in the average number of days of migraine attack presentation per month and comparing the three months before with the three months after treatment administration with two active drugs.
Time Frame: Three months before treatment (Pretreatment), three months after initiating treatment (post-treatment)
Population: It was a straightforward difference between pre and post-treatment in both groups.
Measure: Mean (Standard Deviation); unit: Migraine days by month.
Groups:
- Valproate Group: Comparison between the frequency by month in the three months previous to the starting and the following three months with the use of VPA.
- Memantine: Pretreatment the mean was 5.31 (migraine/days) after treatment was 0.92
Arm/Group | Valproate Group | Memantine
Number analyzed (Participants) | 17 | 16
Migraine days by month.
  Pretreatment | 5.35 (1.11) | 5.31 (1.5)
  Post-treatment | 0.77 (1.16) | 0.93 (1.4)
Statistical Analysis 1: Comparison: Valproate Group vs Memantine; Null hypothesis: Memantine is as effective as valproate in treating episodic migraine; Test type: Non-Inferiority — A new treatment (memantine) that is not much worse or "non-inferior" to the standard treatment (valproate) may be attractive if, compared to it, it is expected to cause fewer side effects or improve quality of life or if its dosing regimen is easier to tolerate; p = 0.9, Wilcoxon (Mann-Whitney) — Comparison between VPA and Memantine was: 0.9 p-value (two-tailed); Memantine 3.534 z corrected for ties 0.0004 p-value (two-tailed) VPA 3.418 z corrected for ties 0.0006 p-value (two-tailed); Mean Difference (Final Values) = 5.3, 95% CI 2-sided [0 to 10], Standard Deviation 14; We made also student t

2. Primary Outcome: The Change in the Intensity of the Pain in a Migraine Attack Will be Measured by a Visual Analogue Scale (VAS).
Description: The possible reduction in the average on the visual analog scale (0-10) comparing three months before and after three months of the treatment with both drugs. We measured both arms of the study.
  0 means without pain. 10 means the worst possible pain in the concept of the patient.
Time Frame: Three months previous and three months after the treatment.
Population: The intensity of pain was measurable by VAS (visual analogous scale) pre and post-treatment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Valproate Group: We pretend to evaluate the difference in the intensity of the pain measurable by the VAS (Visual analogous scale): 0-10 (min to max) pretreatment (8.94 in average) and post-treatment (2.5 in average)
- Memantine: We pretend to evaluate the difference in the Visual Analogue Scale pre (8.5 in average) and posttreatment (4.28 in average)
Arm/Group | Valproate Group | Memantine
Number analyzed (Participants) | 17 | 16
Score on a scale
  Pre-treatment | 8.94 (0.87) | 8.5 (1.36)
  Post-treatment | 2.5 (0.87) | 4.28 (3.65)

3. Primary Outcome: The Migraine Disability Assessment MIDAS Scale Will Measure Before and After the Treatment to Improve the Quality of Life in Both Groups After Three Months of Treatment.
Description: To compare the average of Memantine against the group that receives Valproate before and after starting preventive treatment. Using the Migraine Disability Assessment scale (The score is the sum of days missed from work or school, days of housework missed, days of missed non-work activities, and days of work or school plus days of housework in which productivity in the last three months) to compare punctuation changes. The MIDAS score is divided into four degrees, the minimum score is 0 points, and the maximum score is 70. A higher value represents a higher difficulty to carry out a satisfactory lifestyle, and a score higher than 20 points already represents a high limitation to enjoying daily activities:
  Grade I (0-5 points): Slight limitations and few patient treatment needs. Grade II (6-10 points): Moderate limitations and treatment needs. Grade III (11-20 points) and IV (21 or more points): Severe and significant punctuation treatment needs.
Time Frame: Three months.
Population: MIDAS (Migraine Disability Assessment Score) is a critical evaluation to see the difference between pre and post-treatment with the active drugs we are evaluating.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Valproate Group; Memantine: The incapacity in functionality can be measured by MIDAS (Migraine Disability Assessment)
Arm/Group | Valproate Group | Memantine
Number analyzed (Participants) | 17 | 16
score on a scale
  Pre-treatment | 51.92 (22.67) | 60.87 (15.57)
  Post-treatment | 10.53 (19.97) | 15.57 (14.3)

4. Secondary Outcome: Measure Changes in Weight With the Administration of Active Drugs.
Description: To compare the average weight in both arms before and after Valproate and Memantine administration. The weight will be measured in kilograms, and the initial against the final will be compared.
Time Frame: Three months
Population: Individual weight and mean pre and post-treatment with both drugs.
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Valproate Group: It is well known that VPA can increase the weight of the patient taking this treatment. Therefore, evaluating the patient's status pre and post-treatment is essential.
- Memantine: This is not a common or reported side effect with the use of memantine.
Arm/Group | Valproate Group | Memantine
Number analyzed (Participants) | 17 | 16
kilograms
  Pre-treatment | 71.77 (10.3) | 64.44 (5.8)
  Post-treatment | 72.13 (10.5) | 64.19 (5.3)

5. Other Pre Specified Outcome: To Compare the Adverse Events in the Use of Memantine in Comparision With Valpoate in the Episodic Migraine Treatment.
Description: The number of adverse events and the safety of memantine and valproate. Evaluated according to CTCAE v5.0. There were several side effects, but no one had life-threatening or serious side effects.
Time Frame: Three months
Population: The final analysis was made on a total of 33 participants. However, six left the study because we were in a pandemic situation.
Measure: Count of Participants; unit: Participants
Groups:
- Valproate Group: This is a well know antiepileptic drug with efficacy as a preventive treatment for episodic migraine.
  Besides being an antiepileptic drug, it has been used as a mood stabilizer to prevent episodic migraine.
- Memantine: This is a possible preventive treatment for episodic migraine
  Memantine is a noncompetitive N-methyl-D-aspartate (NMDA) receptor, one of the ionotropic glutamate receptors.
Arm/Group | Valproate Group | Memantine
Number analyzed (Participants) | 17 | 16
Participants
  Somnolence | 6 | 4
  Poor concentration | 0 | 2
  Parasomnia | 1 | 0
  Dizziness | 0 | 2
  No side effects | 10 | 8

ADVERSE EVENTS:
Time Frame: Three months of pretreatment (baseline characteristics) Three months, the duration of the study (12 weeks) Three months post-treatment vigilance.
Groups:
- Valproate Group: VPA is a well know antiepileptic drug with multiple side effects. However, in low doses are a few side effects problems.
- Memantine: Memantine is a tolerable drug. However, it is always necessary to ask for side effects in this type o research.
Arm/Group | Valproate Group | Memantine
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/16
Other Adverse Events (participants affected / at risk) | 7/17 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproate Group (N=17) | Memantine (N=16)
Untoward medical occurrence in the time of study related or not to the drug of the trial (Infections and infestations) | 2 (2) | 1 (1) — Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, in this case, Memantine and valproate.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproate Group (N=17) | Memantine (N=16)
Somnolence (Nervous system disorders) | 6 (6) | 4 (4) — Some participants presented transient somnolence with both drugs without significant problems in the quality of life.
Lack of concentration (Nervous system disorders) | 0 (0) | 2 (2) — Difficult to maintain self-attention and in the environment.
Parasomnia (Nervous system disorders) | 1 (1) | 0 (0) — One of the participants presented parasomnia (nightmare).
dizziness (Nervous system disorders) | 0 (0) | 2 (2) — A transient feeling of instability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT04698525/Prot_003.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT04698525/SAP_005.pdf
  • Informed Consent Form (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT04698525/ICF_002.pdf